CLINICAL TRIAL: NCT04973852
Title: High Intensity Training for Neurological Injury Using Overground Exoskeletons in Inpatient Rehabilitation
Acronym: HIT Exo IP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Shuo-Hsiu Chang, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-21-0262
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury; high intensity; exoskeleton
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Exoskeleton (Experimental): 5 sessions of overground ambulation with wearable exoskeleton where heart rate is monitored over each session.
  Interventions: Device: Ekso

INTERVENTIONS:
Device: Ekso — Exoskeleton walking

SUMMARY:
The purpose of this study is to see if it's possible to reach high cardiovascular intensity training parameters (exercise at a rate that elevates heart rate to the level recommended for improving strength and endurance) while walking in a wearable robotic exoskeleton. This study will also evaluate if exercising at high intensity will lead to improvement in walking ability. Participants in this study will be asked to attend 5 walking training sessions using Ekso exoskeleton. There will be two additional sessions, one before and one after the five training sessions. At these two sessions, study participants will be asked to participate in seated balance, walking speed and endurance tests and breathing assessments.

DETAILED DESCRIPTION:
The purpose of this study is to determine the feasibility and potential efficacy to implement high cardiovascular intensity training parameters (70-80% heart rate reserve) with the use of overground wearable robotic exoskeletons in an inpatient rehabilitation setting for locomotor recovery.

The second aim is to investigate the potential functional improvements in gait after receiving high-intensity locomotor training with an overground exoskeleton, as measured on the 10-meter walk test and six-minute walk test.

ELIGIBILITY:
Inclusion Criteria:

* Able to achieve adequate fit within the exoskeleton
* Diagnosis of CVA or motor incomplete SCI (AIS C or D)
* Sufficient range of motion to attain normal, reciprocal gait pattern, and transition from normal sit to stand or stand to sit
* Intact skin on all surfaces in contact with device and load-bearing surfaces
* Weight <220 pounds

Exclusion Criteria:

* Pregnancy
* Spinal instability
* Unhealed limb or pelvic fractures or any condition restricting weight-bearing in limbs
* Diagnosis of other neurological injuries other than CVA or SCI
* Uncontrolled spasticity (≥3 on Modified Ashworth Scale)
* Colostomy
* Decreased range of motion or contractures in legs (>10° at hips, knees, or ankles)
* Uncontrolled autonomic dysreflexia
* Unresolved deep vein thrombosis
* Inability to tolerate standing due to cardiovascular issues or orthostatic hypotension
* Inability to follow 3 step commands
* Severe comorbidities: active infections, heart, lung, or circulatory conditions
* Pressure sores, impaired skin integrity
* Use of mechanical ventilation for respiratory support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-06 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Heart Rate Reserve Achieved During HIT Gait Training Session while Wearing Exoskeleton | During session 1 (about day 2)
  Heart rate will be monitored continuously and recorded every 5 minutes throughout the session (each session lasts about 60 minutes). Heart rate reserve (HRR) is maximum heart rate (HRmax) minus resting heart rate (HRrest). Target HR ranges will be calculated using age-predicted maximum heart rate (HRmax = 208 - {0.7 * age]) and Karvonen formula (target HRR (70%) = ([0.7 * (HRmax - HRrest)] + HRrest) and (target HRR (80%) = (0.8 * (HRmax - HRrest)] + HRrest). The percentage of HRR achieved during the exoskeleton session is calculated as the percentage of HR readings during the session that are within the 70-80% target HR zone.
Percentage of Heart Rate Reserve Achieved During HIT Gait Training Session | During session 2 (about day 4)
  Heart rate will be monitored continuously and recorded every 5 minutes throughout the session (each session lasts about 60 minutes). Heart rate reserve (HRR) is maximum heart rate (HRmax) minus resting heart rate (HRrest). Target HR ranges will be calculated using age-predicted maximum heart rate (HRmax = 208 - {0.7 * age]) and Karvonen formula (target HRR (70%) = ([0.7 * (HRmax - HRrest)] + HRrest) and (target HRR (80%) = (0.8 * (HRmax - HRrest)] + HRrest). The percentage of HRR achieved during the exoskeleton session is calculated as the percentage of HR readings during the session that are within the 70-80% target HR zone.
Percentage of Heart Rate Reserve Achieved During HIT Gait Training Session | During session 3 (about day 6)
  Heart rate will be monitored continuously and recorded every 5 minutes throughout the session (each session lasts about 60 minutes). Heart rate reserve (HRR) is maximum heart rate (HRmax) minus resting heart rate (HRrest). Target HR ranges will be calculated using age-predicted maximum heart rate (HRmax = 208 - {0.7 * age]) and Karvonen formula (target HRR (70%) = ([0.7 * (HRmax - HRrest)] + HRrest) and (target HRR (80%) = (0.8 * (HRmax - HRrest)] + HRrest). The percentage of HRR achieved during the exoskeleton session is calculated as the percentage of HR readings during the session that are within the 70-80% target HR zone.
Percentage of Heart Rate Reserve Achieved During HIT Gait Training Session | During session 4 (about day 9)
  Heart rate will be monitored continuously and recorded every 5 minutes throughout the session (each session lasts about 60 minutes). Heart rate reserve (HRR) is maximum heart rate (HRmax) minus resting heart rate (HRrest). Target HR ranges will be calculated using age-predicted maximum heart rate (HRmax = 208 - {0.7 * age]) and Karvonen formula (target HRR (70%) = ([0.7 * (HRmax - HRrest)] + HRrest) and (target HRR (80%) = (0.8 * (HRmax - HRrest)] + HRrest). The percentage of HRR achieved during the exoskeleton session is calculated as the percentage of HR readings during the session that are within the 70-80% target HR zone.
Percentage of Heart Rate Reserve Achieved During HIT Gait Training Session | During session 5 (about day 11)
  Heart rate will be monitored continuously and recorded every 5 minutes throughout the session (each session lasts about 60 minutes). Heart rate reserve (HRR) is maximum heart rate (HRmax) minus resting heart rate (HRrest). Target HR ranges will be calculated using age-predicted maximum heart rate (HRmax = 208 - {0.7 * age]) and Karvonen formula (target HRR (70%) = ([0.7 * (HRmax - HRrest)] + HRrest) and (target HRR (80%) = (0.8 * (HRmax - HRrest)] + HRrest). The percentage of HRR achieved during the exoskeleton session is calculated as the percentage of HR readings during the session that are within the 70-80% target HR zone.
Change in Self Selected Gait Speed as Assessed by the 10 Meter Walk Test (10MWT) | Pre Intervention (about 1 day prior to intervention) and 1 Day after session 5 (about day 12)
  During the 10 Meter Walk Test, four marks will be placed on the ground at 0,2,12 and 14 meters. Subjects will walk a total of 14 meters, where the middle 10 meters (between marks 2 and 12 meters) will be timed and recorded as their gait speed. Subjects will complete two attempts at their self-selected pace. The two trials will be averaged and reported as self-selected speed.
Change in Fast Gait Speed as Assessed by the 10 Meter Walk Test (10MWT) | Pre Intervention (about 1 day prior to intervention) and 1 Day after session 5 (about day 12)
  During the 10 Meter Walk Test, four marks will be placed on the ground at 0,2,12 and 14 meters. Subjects will walk a total of 14 meters, where the middle 10 meters (between marks 2 and 12 meters) will be timed and recorded as their gait speed. Subjects will complete two attempts at their fastest pace. The two trials will be averaged and reported as fast gait speed.
Change in Walking Endurance as Assessed by the 6 Minute Walk Test (6MWT) | Pre Intervention (about 1 day prior to intervention) and 1 Day after session 5 (about day 12)
  The 6 Minute Walk Test will measure the distance subjects can walk over six minutes. Subjects will walk along a 100-foot hallway as many times as they can in 6 minutes. Subjects are allowed to rest as needed; however, the timer continues to run for 6 minutes consecutively, whether they are standing or walking.

SECONDARY OUTCOMES:
Change in Seated Dynamic Reach as Assessed by the Modified Functional Reach Test | Pre Intervention (about 1 day prior to intervention) and 1 Day after session 5 (about day 12)
  The Modified Functional Reach Test measures the maximum distance an individual can reach forward from a seated position. This will be reported as an average of three trials.
Change in Spatial-Temporal Gait Parameters as assessed by the GAITRite pressure map (step length parameter) | Pre Intervention (about 1 day prior to intervention) and 1 Day after session 5 (about day 12)
  The GAITRite pressure map will be used during the 10MWT. This pressure map will digitally record the subject's footprints' placement and pressure as they walk over it during the 10MWT. This assessment will indicate several temporospatial gait parameters. The average step length (measured in centimeters) will be reported.
Change in Spatial-Temporal Gait Parameters as assessed by the GAITRite pressure map (stride length parameter) | Pre Intervention (about 1 day prior to intervention) and 1 Day after session 5 (about day 12)
  The GAITRite pressure map will be used during the 10MWT. This pressure map will digitally record the subject's footprints' placement and pressure as they walk over it during the 10MWT. This assessment will indicate several temporospatial gait parameters. The average stride length (measured in centimeters) will be reported.
Change in Spatial-Temporal Gait Parameters as assessed by the GAITRite pressure map (single support parameter) | Pre Intervention (about 1 day prior to intervention) and 1 Day after session 5 (about day 12)
  The GAITRite pressure map will be used during the 10MWT. This pressure map will digitally record the subject's footprints' placement and pressure as they walk over it during the 10MWT. This assessment will indicate several temporospatial gait parameters. The average time spent in single limb support (measured as percentage of total gait cycle) will be reported.
Change in Spatial-Temporal Gait Parameters as assessed by the GAITRite pressure map (double support parameter) | Pre Intervention (about 1 day prior to intervention) and 1 Day after session 5 (about day 12)
  The GAITRite pressure map will be used during the 10MWT. This pressure map will digitally record the subject's footprints' placement and pressure as they walk over it during the 10MWT. This assessment will indicate several temporospatial gait parameters. The average time spent in double limb support (measured as percentage of total gait cycle) will be reported.
Change in Spatial-Temporal Gait Parameters as assessed by the GAITRite pressure map (swing time parameter) | Pre Intervention (about 1 day prior to intervention) and 1 Day after session 5 (about day 12)
  The GAITRite pressure map will be used during the 10MWT. This pressure map will digitally record the subject's footprints' placement and pressure as they walk over it during the 10MWT. This assessment will indicate several temporospatial gait parameters. The average time spent in swing phase (measured as percentage of total gait cycle) will be reported.
Change in Spatial-Temporal Gait Parameters as assessed by the GAITRite pressure map (stance time parameter) | Pre Intervention (about 1 day prior to intervention) and 1 Day after session 5 (about day 12)
  The GAITRite pressure map will be used during the 10MWT. This pressure map will digitally record the subject's footprints' placement and pressure as they walk over it during the 10MWT. This assessment will indicate several temporospatial gait parameters. The average time spent in stance phase (measured as percentage of total gait cycle) will be reported.
Change in Spatial-Temporal Gait Parameters as assessed by the GAITRite pressure map (heel to heel base of support time parameter) | Pre Intervention (about 1 day prior to intervention) and 1 Day after session 5 (about day 12)
  The GAITRite pressure map will be used during the 10MWT. This pressure map will digitally record the subject's footprints' placement and pressure as they walk over it during the 10MWT. This assessment will indicate several temporospatial gait parameters. The average heel to heel base of support (measured in centimeters) will be reported.
Change in Metabolic Expenditure during 10MWT, as Assessed by Oxygen Consumption | Pre Intervention (about 1 day prior to intervention) and 1 Day after session 5 (about day 12)
  Change in metabolic expenditure during 10MWT will be indicated by energy expenditure. Energy Expenditure will be measured by the K4 b2 Cosmed as follows: Oxygen cost will be calculated from oxygen consumption as the product of gait speed and body weight. Oxygen consumption will be collected on a breath-by-breath basis measured by a portable metabolic system (K4 b2 Cosmed). Prior to the testing, the system will be calibrated using room air and reference gas mixture. During the testing, the subject will wear a face mask and a heart rate monitor at all times and will be asked to breathe normally. The average oxygen cost will be reported as VO2 peak during 10MWT.
Change in Metabolic Expenditure during 6MWT, as Assessed by Oxygen Consumption | Pre Intervention (about 1 day prior to intervention) and 1 Day after session 5 (about day 12)
  Change in metabolic expenditure during 6MWT will be indicated by energy expenditure. Energy Expenditure will be measured by the K4 b2 Cosmed as follows: Oxygen cost will be calculated from oxygen consumption as the product of gait speed and body weight. Oxygen consumption will be collected on a breath-by-breath basis measured by a portable metabolic system (K4 b2 Cosmed). Prior to the testing, the system will be calibrated using room air and reference gas mixture. During the testing, the subject will wear a face mask and a heart rate monitor at all times and will be asked to breathe normally. The average oxygen cost will be reported as VO2 peak during 6MWT.

CONTACTS AND LOCATIONS:
Overall Officials: Shuo-Hsiu (James) Chang, Principal Investigator — The University of Texas Health Sciences Center at Houston
Locations (1):
- NeuroRecovery Research Center at TIRR Memorial Hermann, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brazg G, Fahey M, Holleran CL, Connolly M, Woodward J, Hennessy PW, Schmit BD, Hornby TG. Effects of Training Intensity on Locomotor Performance in Individuals With Chronic Spinal Cord Injury: A Randomized Crossover Study. Neurorehabil Neural Repair. 2017 Oct-Nov;31(10-11):944-954. doi: 10.1177/1545968317731538. Epub 2017 Oct 30. PMID 29081250
- [Background] Lotter JK, Henderson CE, Plawecki A, Holthus ME, Lucas EH, Ardestani MM, Schmit BD, Hornby TG. Task-Specific Versus Impairment-Based Training on Locomotor Performance in Individuals With Chronic Spinal Cord Injury: A Randomized Crossover Study. Neurorehabil Neural Repair. 2020 Jul;34(7):627-639. doi: 10.1177/1545968320927384. Epub 2020 Jun 1. PMID 32476619
- [Background] Hornby TG, Henderson CE, Plawecki A, Lucas E, Lotter J, Holthus M, Brazg G, Fahey M, Woodward J, Ardestani M, Roth EJ. Contributions of Stepping Intensity and Variability to Mobility in Individuals Poststroke. Stroke. 2019 Sep;50(9):2492-2499. doi: 10.1161/STROKEAHA.119.026254. Epub 2019 Aug 22. PMID 31434543
- [Background] Holleran CL, Rodriguez KS, Echauz A, Leech KA, Hornby TG. Potential contributions of training intensity on locomotor performance in individuals with chronic stroke. J Neurol Phys Ther. 2015 Apr;39(2):95-102. doi: 10.1097/NPT.0000000000000077. PMID 25784587
- [Background] Holleran CL, Straube DD, Kinnaird CR, Leddy AL, Hornby TG. Feasibility and potential efficacy of high-intensity stepping training in variable contexts in subacute and chronic stroke. Neurorehabil Neural Repair. 2014 Sep;28(7):643-51. doi: 10.1177/1545968314521001. Epub 2014 Feb 10. PMID 24515925
- [Background] Moore JL, Nordvik JE, Erichsen A, Rosseland I, Bo E, Hornby TG; FIRST-Oslo Team. Implementation of High-Intensity Stepping Training During Inpatient Stroke Rehabilitation Improves Functional Outcomes. Stroke. 2020 Feb;51(2):563-570. doi: 10.1161/STROKEAHA.119.027450. Epub 2019 Dec 30. PMID 31884902
- [Background] Leech KA, Hornby TG. High-Intensity Locomotor Exercise Increases Brain-Derived Neurotrophic Factor in Individuals with Incomplete Spinal Cord Injury. J Neurotrauma. 2017 Mar 15;34(6):1240-1248. doi: 10.1089/neu.2016.4532. Epub 2017 Jan 18. PMID 27526567
- [Background] Hornby TG, Holleran CL, Hennessy PW, Leddy AL, Connolly M, Camardo J, Woodward J, Mahtani G, Lovell L, Roth EJ. Variable Intensive Early Walking Poststroke (VIEWS): A Randomized Controlled Trial. Neurorehabil Neural Repair. 2016 Jun;30(5):440-50. doi: 10.1177/1545968315604396. Epub 2015 Sep 3. PMID 26338433
- [Background] Holleran CL, Hennessey PW, Leddy AL, Mahtani GB, Brazg G, Schmit BD, Hornby TG. High-Intensity Variable Stepping Training in Patients With Motor Incomplete Spinal Cord Injury: A Case Series. J Neurol Phys Ther. 2018 Apr;42(2):94-101. doi: 10.1097/NPT.0000000000000217. PMID 29547484